CLINICAL TRIAL: NCT05724082
Title: The Effect of Household Air Pollution on Lung Function Growth in Infants With Pneumonia in Sub-Saharan Africa
Acronym: PLUS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Peter Moschovis, Principal Investigator, Pediatric Pulmonologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2019P000649
Record Dates: First submitted 2022-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pneumonia; Pollution; Exposure; Lung Function Decreased; Chronic Respiratory Disease; Pediatric Respiratory Diseases; Lungs; Developmental Disorder
MeSH Terms: conditions — Pneumonia; Respiratory Insufficiency; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The air filtration system will be cycled monthly, with active filtration alternating with no filtration for one month on/one month off.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clean air intervention (Experimental): See detailed description
  Interventions: Other: Clean Air Intervention

INTERVENTIONS:
Other: Clean Air Intervention — Based on findings from preliminary focus groups/in-depth interviews, staff will introduce various components of established clean air interventions to each household. Each household will receive interventions, depending on their known risk factors, exposures, and willingness to trial the intervention.
  Study staff will ask the primary cook to complete a time-activity diary during the intervention period that includes cooking episodes, duration of cooking, stove(s) used, type of food cooked, and number of people for whom the meal was cooked. Staff will continuously monitor use of the LPG/pellet stove and any other stoves owned by the household with the Berkeley Stove Use Monitoring System, a temperature logger attached to the stove to quantify the number of stove uses / time of use . Study staff will use similar loggers to monitor use of other devices installed including the air purifiers, lighting etc.

SUMMARY:
This study will evaluate the feasibility and acceptability of a household-based clean air intervention

DETAILED DESCRIPTION:
A clean air intervention will be implemented in each household, including HEPA- based air filtration, solar lighting, and education. The air filtration system will be cycled monthly, with active filtration alternating with no filtration for one month on/one month off. To determine the effect of the clean air intervention within the household, PM2.5 concentration during each cycle and lung function will be measured among household members.

ELIGIBILITY:
Inclusion Criteria:

* Age < 12 months

  • First episode of WHO-defined severe pneumonia22: cough or difficulty breathing with
* Oxygen saturation < 90% or central cyanosis,
* Severe respiratory distress, or
* Signs of pneumonia with a general danger sign
* Be willing to commit to entire 2 years of follow up visits.
* (Controls) Matched to each case on age (+/-1 month), sex, and community

Exclusion Criteria:

* Craniofacial, cardiac or other major malformation
* Neuromuscular condition that affects respiration
* Outside Smart Discharges Project catchment area
* Prior hospitalizations or known episodes of respiratory illness or episodes of pneumonia before index admission,

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the clean intervention | 2 years
  Adherence with the intervention (% total up-time of the air purifier)

SECONDARY OUTCOMES:
Air quality | Up to 2 years
  PM2.5 concentration
Pulmonary function testing | Up to 2 years
  Pulmonary function testing will be performed in household members
Acceptability of using air filter device | Up to 2 years
  Acceptability will be assessed using structured interviews with participating households.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Moschovis, MD, Principal Investigator — Massachusetts General Hospital; Jerome Kabakyenga, MBChB, MPH, PhD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No